CLINICAL TRIAL: NCT06404788
Title: Anxiety Level Among Polish Patients With Chronic Low Back Pain: a Cross-sectional Study
Brief Title: Anxiety Level Among Patients With Chronic Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Tomasz Jurys (Other)
Responsible Party: Sponsor-Investigator, Tomasz Jurys, PhD, University Lecturer, Medical University of Silesia
Organization: Medical University of Silesia (Other)
Other Study IDs: BNW/NWN/0052/KB/97/24
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Anxiety Disorders; Anxiety Disorders and Symptoms; Lower Back Pain; Chronic Pain
Keywords: chronic pain; low back pain; anxiety
MeSH Terms: conditions — Anxiety Disorders; Low Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cross-sectional study is to learn about the intensity of anxiety symptoms among Polish people suffering from chronic lower back pain. The main question it aims to answer is:

What is the severity of anxiety symptoms among the Polish population of patients suffering from chronic lower back pain?

ELIGIBILITY:
Inclusion Criteria:

* age minimum 18 years old
* chronic low back pain (duration longer than 3 months)
* native Polish speaker
* people who gave informed consent to participate in the study

Exclusion Criteria:

* trauma/ surgery on the low back within the past one year
* diagnosis of severe mental illness
* pregnant within the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult people with chronic low back pain waiting for consultation or physiotherpay intervention in primary care clinic or physiotherapy clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Severity | up to 10 months
  Severity of the anxiety symptoms

IPD SHARING:
Plan to Share IPD: No